CLINICAL TRIAL: NCT02883088
Title: Relationship Between Coronary Plaque Morphology of Left Anterior Descending Artery and Long Term Clinical Outcome: the CLIMA Study
Brief Title: Relationship Between OCT Coronary Plaque Morphology and Clinical Outcome
Acronym: CLIMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: San Giovanni Addolorata Hospital (Other)
Collaborators: Centro per la Lotta Contro l'Infarto - Fondazione Onlus (Other)
Responsible Party: Principal Investigator, Francesco Prati, Dr., San Giovanni Addolorata Hospital
Other Study IDs: CLI-01-2013
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: Optical coherence tomograhpy; registry; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAD-group: Subjects over 18 years who are undergoing Frequency Domain - Optical Coherence Tomography (FD-OCT) evaluation of the native left anterior descending artery during clinically indicated coronary angiography regardless of the clinical syndrome (silent ischemia, effort angina or acute coronary syndrome).
  Interventions: Procedure: Frequency Domain - Optical Coherence Tomography (FD-OCT)

INTERVENTIONS:
Procedure: Frequency Domain - Optical Coherence Tomography (FD-OCT) — FD-OCT assessment of the native proximal-mid left descending artery during clinically indicated coronary angiography

SUMMARY:
The multicenter observational CLIMA registry has been conceived to explore correlation between OCT morphology of atherosclerotic plaques located in the left anterior descending artery with mid and long term clinical outcome.

DETAILED DESCRIPTION:
Acute myocardial infarction (MI) is commonly caused by plaque ulceration and subsequent local thrombosis. Plaques that tend to rupture are typically characterized by a large superficial lipid pool, delimited by a thin fibrous cap and often exhibit local signs of inflammation. Such atherosclerotic lesions are commonly described as vulnerable plaques (1-4).

Identification of these plaque features with imaging modalities is potentially a valid approach to identify patients at increased risk of M (5). Optical coherence tomography is capable of visualizing superficial plaque components at a high resolution (in the range of 10-15 microns) and can depict all the features of plaque vulnerability or thrombogenicity (6,7).

The aim of the study is to relate presence of multiple OCT criteria of plaque vulnerability with following clinical events in a subset of coronary lesions. For this purpose all plaques in the proximal-mid portion of the left anterior descending artery will be evaluated with FD-OCT assessing the following criteria:

* minimum lumen area (MLA) <3.5 mm2:
* fibrous cap minimum thickness <75 µm:
* lipid arc extension >180°;
* presence of macrophages;

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Patients with clinical indication to coronary angiography undergoing OCT evaluation of the left anterior descending artery regardless of the clinical syndrome;
* Patients with at least 30 mm of naïve OCT-assessable proximal-mid left anterior descending artery;
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent to the procedure;

Exclusion Criteria:

* Female with childbearing potential or lactating;
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Advanced heart failure (NYHA III-IV)
* Previous Coronary artery by-pass surgery
* Previous stenting of proximal-mid left anterior descending artery with residual untreated segment <30mm.
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study;
* Heavily calcified vessel and/or lesion which cannot be successfully imaged by OCT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive subjects undergoing OCT assessment of the proximal left descending artery coronary during coronary angiography should be screened for eligibility.
  Patients will be enrolled from participating centers at the time of OCT assessment and prospectively investigated to evaluate clinical outcome.
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1-year
  Composite of cardiac death and/or target vessel myocadial infarction

SECONDARY OUTCOMES:
Major adverse cardiac events | 3-year
  Composite of cardiac death and/or target vessel myocadial infarction

OTHER OUTCOMES:
Predictive value of single OCT criteria of plaque vulnerability | 1-year and 3-year
  Predictive value of minimum lumen area, fibrous cap thickness, lipid arc extension, presence of macrophages at the explored plaques

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Prati, MD, Principal Investigator — San Giovanni Addolorata Hospital
Locations (14):
- Italy (12):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Ospedale Brotzu, Cagliari
  - Presidio Ospedaliero Sant'Elia, Caltanissetta
  - University of Catania, Catania
  - GVM Care and Research, E. S. Health Science Foundation, Cotignola
  - Misericordia Hospital, Grosseto
  - Ospedale Civile Ferdinando Veneziale, Isernia
  - Policlinico G. Martino, Messina
  - Centro Cardiologico Monzino IRCCS, Milan
  - San Giovanni-Addolorata Hospital, Rome
  - Università Cattolica Del Sacro Cuore, Rome
  - Presidio Ospedaliero Umberto I°, Syracuse
- Central Clinical Hospital of the Ministry of Interior, Warsaw, Poland
- Hospital Universitario Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falk E, Shah PK, Fuster V. Coronary plaque disruption. Circulation. 1995 Aug 1;92(3):657-71. doi: 10.1161/01.cir.92.3.657. No abstract available. PMID 7634481
- [Background] De Caterina R. Endothelial dysfunctions: common denominators in vascular disease. Curr Opin Clin Nutr Metab Care. 2000 Nov;3(6):453-67. doi: 10.1097/00075197-200011000-00007. PMID 11085831
- [Background] Naghavi M, Libby P, Falk E, Casscells SW, Litovsky S, Rumberger J, Badimon JJ, Stefanadis C, Moreno P, Pasterkamp G, Fayad Z, Stone PH, Waxman S, Raggi P, Madjid M, Zarrabi A, Burke A, Yuan C, Fitzgerald PJ, Siscovick DS, de Korte CL, Aikawa M, Juhani Airaksinen KE, Assmann G, Becker CR, Chesebro JH, Farb A, Galis ZS, Jackson C, Jang IK, Koenig W, Lodder RA, March K, Demirovic J, Navab M, Priori SG, Rekhter MD, Bahr R, Grundy SM, Mehran R, Colombo A, Boerwinkle E, Ballantyne C, Insull W Jr, Schwartz RS, Vogel R, Serruys PW, Hansson GK, Faxon DP, Kaul S, Drexler H, Greenland P, Muller JE, Virmani R, Ridker PM, Zipes DP, Shah PK, Willerson JT. From vulnerable plaque to vulnerable patient: a call for new definitions and risk assessment strategies: Part I. Circulation. 2003 Oct 7;108(14):1664-72. doi: 10.1161/01.CIR.0000087480.94275.97. PMID 14530185
- [Background] Narula J, Nakano M, Virmani R, Kolodgie FD, Petersen R, Newcomb R, Malik S, Fuster V, Finn AV. Histopathologic characteristics of atherosclerotic coronary disease and implications of the findings for the invasive and noninvasive detection of vulnerable plaques. J Am Coll Cardiol. 2013 Mar 12;61(10):1041-51. doi: 10.1016/j.jacc.2012.10.054. PMID 23473409
- [Background] Jang IK, Bouma BE, Kang DH, Park SJ, Park SW, Seung KB, Choi KB, Shishkov M, Schlendorf K, Pomerantsev E, Houser SL, Aretz HT, Tearney GJ. Visualization of coronary atherosclerotic plaques in patients using optical coherence tomography: comparison with intravascular ultrasound. J Am Coll Cardiol. 2002 Feb 20;39(4):604-9. doi: 10.1016/s0735-1097(01)01799-5. PMID 11849858
- [Background] Jang IK, Tearney GJ, MacNeill B, Takano M, Moselewski F, Iftima N, Shishkov M, Houser S, Aretz HT, Halpern EF, Bouma BE. In vivo characterization of coronary atherosclerotic plaque by use of optical coherence tomography. Circulation. 2005 Mar 29;111(12):1551-5. doi: 10.1161/01.CIR.0000159354.43778.69. Epub 2005 Mar 21. PMID 15781733
- [Background] Kawasaki M, Bouma BE, Bressner J, Houser SL, Nadkarni SK, MacNeill BD, Jang IK, Fujiwara H, Tearney GJ. Diagnostic accuracy of optical coherence tomography and integrated backscatter intravascular ultrasound images for tissue characterization of human coronary plaques. J Am Coll Cardiol. 2006 Jul 4;48(1):81-8. doi: 10.1016/j.jacc.2006.02.062. Epub 2006 Jun 9. PMID 16814652
- [Derived] Biccire FG, Fabbiocchi F, Gatto L, La Manna A, Ozaki Y, Romagnoli E, Marco V, Boi A, Fineschi M, Piedimonte G, Cerrato E, Musto C, Taglieri N, Di Giorgio A, Vizzari G, Ruscica G, Canova PA, Vergallo R, Burzotta F, Limbruno U, Albertucci M, Raber L, Crea F, Alfonso F, Arbustini E, Stone GW, Prati F. Long-Term Prognostic Impact of OCT-Derived High-Risk Plaque Features: Extended Follow-Up of the CLIMA Study. JACC Cardiovasc Interv. 2025 Jun 9;18(11):1361-1372. doi: 10.1016/j.jcin.2025.04.044. PMID 40500004
- [Derived] Budassi S, Biccire FG, Gatto L, Scorza M, Marco V, Porta Y, Sammartini E, Paoletti G, Debelak C, Di Pietro R, Circhetta S, Albertucci M, Burzotta F, Ozaki Y, Canova PA, Piedimonte G, Alfonso F, Arbustini E, Prati F. Independent role of atherosclerotic plaque composition and extension in predicting the risk of cardiac events: a CLIMA substudy. Int J Cardiovasc Imaging. 2024 Dec;40(12):2535-2543. doi: 10.1007/s10554-024-03260-2. Epub 2024 Oct 21. PMID 39432135
- [Derived] Biccire FG, Debelak C, Varricchione G, Budassi S, Gatto L, Romagnoli E, Di Pietro R, Sammartini E, Marco V, Paoletti G, Burzotta F, Ozaki Y, Pastori D, Alfonso F, Arbustini E, Prati F. Sex-specific features of optical coherence tomography detected plaque vulnerability related to clinical outcomes: insights from the CLIMA study. Int J Cardiovasc Imaging. 2023 Apr;39(4):873-881. doi: 10.1007/s10554-022-02775-w. Epub 2022 Dec 19. PMID 36534217